CLINICAL TRIAL: NCT04156958
Title: An Exploratory Study to Evaluate Efficacy and Safety of Fruquintinib as Second-line Treatment for Patients With Advanced or Metastatic Biliary Tract Cancer
Brief Title: Fruquintinib as Second-line Treatment for Advanced/Metastatic Biliary Tract Adenocarcinoma
Acronym: FSTAMBTA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2165
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Biliary Tract Adenocarcinoma
Keywords: biliary tract adenocarcinoma; fruquintinib; anti-angiogenesis
MeSH Terms: interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib Arm (Other): Fruquintinib, 5 mg once daily for 21 days, followed by 7 days off (28 days/cycle) treatment until progression, unacceptable toxicity, or withdrawal unless toxicity not relieved after dose adjustment.
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib will be administered orally at a dose of 5 mg/d, 3 weeks on, 1 week off (4 weeks as a cycle) until progression, unacceptable toxicity, or withdrawal unless toxicity not relieved after dose adjustment.
  Other Names: Elunate

SUMMARY:
The prospective, multicenter, single-arm design study is to evaluate the efficacy and safety of fruquintinib for patients with advanced or metastatic biliary tract adenocarcinoma who failed first-line chemotherapy with gemcitabine, platinum/S-1, and albumin paclitaxel.

DETAILED DESCRIPTION:
Biliary tract cancer arises from the epithelial cells of the bile ducts. Until nowadays, no standard second-line treatment has been established following recurrence from the first-line treatment. Angiogenesis plays a key role in the carcinogenesis and development of biliary tract adenocarcinoma. Studies have shown that VEGF is expressed in more than 50% of biliary tract adenocarcinoma, and microvessel density is significantly associated with tumor progression, metastasis, and prognosis. Fruquintinib (trade name: Elunate) is a novel small molecule tyrosine kinase inhibitor. It is currently being evaluated in clinical trials for multiple cancers including lung cancer, gastric cancer and colorectal cancer and showed strong anti-tumor activity. The aim of the study is to evaluate the efficacy and safety of fruquintinib for patients with advanced or metastatic biliary tract adenocarcinoma who failed first-line chemotherapy.

The trial is a prospective, multicenter, single-arm design study. Eligible participants with advanced or metastatic biliary tract adenocarcinoma who have failed first-line chemotherapy with gemcitabine, platinum/S-1, and albumin paclitaxel. The study will explore the efficacy and safety of second-line treatment with fruquintinib, and quality of life during treatment. Tumor assessment was performed every 8 weeks as defined by RECIST 1.1. Blood samples will be collected at baseline (before treatment) and 2 weeks after treatment, and cfDNA will be collected for gene detection analysis to evaluate the correlation between different gene mutations and their changes and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* （1） Patients must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.

  （2） Age ≥18 years. （3） Histologically or cytologically confirmed diagnosis of advanced or metastatic biliary tract adenocarcinoma （4） First-line chemotherapy failed (tumor progression or intolerable adverse events).

  （5） The expected survival is no less than 3 months. （6） ECOG PS≤1. （7） At least one measurable lesion according to RECIST 1.1 criteria. （8） Adequate organ function including the following:
  * Total bilirubin ≤3 times upper limit of normal (ULN),
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤5×ULN,
  * Alkaline phosphatase≤2.5×ULN (If the tumor invaded the liver, ≤5×ULN),
  * Serum creatinine≤1.5×ULN,
  * Serum amylase and lipase≤1.5×ULN,
  * International standardized ratio (INR)/partial prothrombin time (PTT)≤1.5×ULN;
  * Platelet count ≥ 75,000 /mm3.
  * Hemoglobin (Hb) ≥ 9 g/dL.
  * Absolute neutrophil count (ANC) ≥ 1500/mm3. （9） Strict contraception.

Exclusion Criteria:

* （1） Unable to comply with the research program or procedures. （2） Undergoing other drug clinical trials, or has participated in any drug clinical trials one month before enrollment.

  （3） Uncontrolled hypertension (systolic pressure ≥140 mm Hg or diastolic pressure ≥ 90 mm Hg on repeated measurement) despite optimal medical management.

  （4） Active or clinically significant cardiac disease:
  * Congestive heart failure > New York Heart Association (NYHA ) class 2;
  * Active coronary artery disease;
  * Arrhythmias requiring treatment other than β-blocker or digoxin;
  * Unstable angina (with angina symptoms at rest), new angina within 3 months before enrollment, or new myocardial infarction within 6 months before enrollment （5） Evidence or history of bleeding diathesis or coagulopathy. （6） Grade 3 bleeding events 4 weeks before enrollment. （7） Thromboembolism or arteriovenous events, such as cerebrovascular events (including transient ischemic attack), deep vein thrombosis or pulmonary embolism, occurred 6 months before enrollment.

    （8） Currently taking anticoagulants. （9） Other tumors that have not been treated or exist at the same time, except carcinoma in situ of the cervix, treated basal cell carcinoma or superficial bladder tumor. If the tumor has been cured and no evidence of disease has been found for more than 3 years, the patient can be enrolled. All other tumors must be treated at least 3 years before enrollment.

    （10） Patients with pheochromocytoma. （11） Patients with a history of HIV infection or active hepatitis B/C. （12） Ongoing > level 2 infection. （13） Symptomatic brain metastasis or meningioma. （14） Unhealed wounds, ulcers or fractures. （15） Renal failure patients requiring blood or peritoneal dialysis. （16） Dehydration≥ 1 grade （17） Epileptic that need medication （18） Proteinuria≥ 3 grade (Urinary protein > 3.5g / 24hour) （19） Active, symptomatic interstitial pneumonia, pleural or ascites that causes dyspnea (dyspnea ≥ 2 grade) （20） History of organ transplantation. (including corneal transplantation). （21） Allergic to research drugs or similar drugs, or suspected allergies. （22） Malabsorption patients. （23） Pregnant or lactating women. （24） Investigator believes that patients who are not suitable for the study. （25） Medical, psychological or social conditions can affect the recruitment of patients and evaluation for study results.

    （26） Other anti-tumor therapy (chemotherapy, radiotherapy, surgery, immunotherapy, biotherapy, chemoembolization) other than investigator drugs (fruquintinib). Palliative external irradiation for non-target lesions is allowed.

    （27） Previously used fruquintinib or other angiogenesis inhibitors. （28） Major surgery 4 weeks before recruitment, open biopsy or major trauma surgery. (excluding biliary stents, or percutaneous biliary drainage) （29） Treatment with anti-tumor Chinese herbal medicine. （30） History of allogeneic blood transfusion within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to 5 years
  Defined as the time from the date of enrollment to the first date of documented objective progression disease or of death from any cause

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 5 years
  Defined as the percentage of patients who have a partial or complete response to therapy
Disease control rate (DCR) | Up to 5 years
  Defined as the percentage of patients who have achieved complete response, partial response and stable disease
Overall survival (OS) | Up to 5 years
  Defined as the time from the date of enrollment to the date of death from any cause
Safety and Tolerability | 3 months after the last administration of fruquintinib
  Defined by treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Qiu Li, M.D., Principal Investigator — West China Hospital
Locations (7):
- China (7):
  - Chinese PLA General Hospital 5th Medical Center, Beijing, Beijing Municipality
  - Hebei Tumor Hospital, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No